CLINICAL TRIAL: NCT05338372
Title: Forest Therapy on Physical and Psychological Parameters in the General Population
Brief Title: Effects of Forest Therapy on Physical and Psychological Parameters in the General Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Andreas Michalsen, Prof. Dr. Andreas Michalsen, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KWT1
Record Dates: First submitted 2022-04-11; First posted 2022-04-21 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: General Population
MeSH Terms: interventions — Forest Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Two days forest therapy (Experimental)
  Interventions: Behavioral: Two days forest therapy
- Three days forest therapy (Experimental)
  Interventions: Behavioral: Three days forest therapy

INTERVENTIONS:
Behavioral: Two days forest therapy — Participants attend two days (with a break day in between) of two-hour forest therapy at the Friedrichsruh, Barntrup or Wernigerode sites, led by an INFTA-certified forest therapy guide.
  Arms: Two days forest therapy
Behavioral: Three days forest therapy — Participants attend three days of two-hour forest therapy at the Friedrichsruh, Barntrup or Wernigerode sites, led by an INFTA-certified forest therapy guide.
  Arms: Three days forest therapy

SUMMARY:
In recent years, nature and forest therapy has increasingly become the focus of medical research. Recent scientific findings indicate overall positive effects of nature and forest therapy on physical and mental health. In Asia and Australia, it has already been implemented as a public health concept of prevention and health promotion. The aim of the project is to replicate the experience gained in Asia over the last three decades on the physical and psychological effects of nature/forest therapy in the context of the German forest and to investigate it further scientifically.

ELIGIBILITY:
Inclusion criteria:

* Women and men aged 18 to 90 years.
* Capacity to consent

Exclusion criteria:

* Serious acute or chronic medical conditions
* Immobility or limitation of mobility due to orthopedic, neurological or other medical causes
* Participation in another study
* Serious mental illness
* Pregnancy and lactation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2022-06-04 (Actual); Study Completion 2022-06-04 (Actual)

PRIMARY OUTCOMES:
Profile of Mood States (POMS) | Change from baseline POMS score at 3 days
  Assessing full scale, range 1-7, lower score meaning a better outcome

SECONDARY OUTCOMES:
Perceived Benefits of Nature Questionnaire (PBNQ) | Change from baseline PBNQ score at 3 days
  Assessing full scale, range 1-7, lower score meaning a better outcome
Subjective Vitality Scale state (SVS-G state) | Change from baseline SVS-G score at 3 days
  Assessing full scale, range 1-80, higher score meaning a better outcome
Complaint List (B-LR) | Change from baseline B-LR score at 3 days
  Assessing full scale, range 1-50, lower score meaning a better outcome
Perceive Stress Questionaire (PSQ) | Change from baseline PSQ score at 3 days
  Assessing full scale, range 1-40, lower score meaning a better outcome
State-Trait Anxiety Inventory (STAI) | Change from baseline STAI score at 3 days
  Assessing state anxiety. The scale ranges from 1 to 8. Higher scores correspond to higher levels of anxiety (after recoding three inverted items).
PROMIS Scale v1.2 - Global Health | Change from baseline PROMIS score at 3 days
  The scale ranges from 1 to 5, where 1 is the lowest level and 5 is the highest level. Higher scores reflect better functioning.
Allgemeine Selbstwirksamkeit Kurzskala (ASKU) | Change from baseline ASKU score at 3 days
  Assessing full scale, the scale ranges from 1 to 5. Higher scores correspond to better outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Charite University, Berlin, Germany